CLINICAL TRIAL: NCT01279629
Title: Open Clinical Study, Comparing Non-inferiority for Efficacy of the Drug Tazarotene 0.1% Versus the Comparator Drug Calcipotriol 0.005% in the Treatment of Chronic Plaque Psoriasis
Brief Title: Open Clinical Study, Comparing Non-inferiority of Chronic Plaque Psoriasis
Acronym: MED
Status: Suspended | Type: Observational
Sponsor: Glenmark Farmacêutica Ltda (Industry)
Responsible Party: Glenmark Farmacêutica Ltda, Glenmark Farmacêutica Ltda
Other Study IDs: MED 865-10v3
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-01

CONDITIONS: Plaque Psoriasis
Keywords: chronic plaque psoriasis; To evaluate the efficacy of the drugs under study for treating chronic plaque psoriasis
MeSH Terms: interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tazarotene 0.1%
  Interventions: Drug: Each patient will receive a sample of the drug test (tazarotene 0.1%) and a control sample of the drug (calcipotriene 0.005%).
- Calcipotriol 0.005%
  Interventions: Drug: Each patient will receive a sample of the drug test (tazarotene 0.1%) and a control sample of the drug (calcipotriene 0.005%).

INTERVENTIONS:
Drug: Each patient will receive a sample of the drug test (tazarotene 0.1%) and a control sample of the drug (calcipotriene 0.005%). — Apply the medication once daily, preferably at night, in quantities sufficient to cover only the lesions with a thin layer of the product (an average of 2 mg/cm2).Apply only in lesions of the right hemisphere.

SUMMARY:
The purpose of this study is:

To evaluate the efficacy of the drugs under study for treating chronic plaque psoriasis.

- Population:

50 patients will be selected from both sexes, healthy, between 18 and 65 years with a clinical diagnosis of chronic plaque psoriasis with PASI <20%, according to the criteria of inclusion and exclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Between 18 and 65
* A patient with chronic plaque psoriasis
* PASI <20%
* Presence of bilateral lesions with at least 2 cm in diameter and each with some degree of symmetry
* Levels of serum calcium and phosphorus within the normal range of reference or in case of changes, classified as irrelevant by the investigator
* In the case of female patients, agreement or maintenance of safe use of contraception such as barrier (condom, diaphragm), hormonal contraceptives (pills, implants or injections), IUDs, or abstinence (no sex)
* Reading, understanding, agreement and signature of the patient in the Term of Consent.

Exclusion Criteria:

* Gestation (confirmed by urine test indicator)
* Lactation
* History of hypersensitivity to components of medicines
* Psoriasis with different clinical presentation of the plates
* Clinical picture of psoriasis involving only the scalp, face, groin, armpit and / or other intertriginous area
* Patient requires the use of concomitant medication (topical or systemic) that may alter the course of the disease during the study period
* Use of any systemic treatment for psoriasis within 12 weeks before the start of the study
* Use of systemic corticosteroids within 28 days before the start of the study
* Use of topical corticosteroids or other topical therapies in the areas of assessment within 02 weeks before the start of the study
* Use of phototherapy (UVB / UVA-P) within 04 weeks before the start of the study
* Patients who have participated in another clinical study within 30 days before the start of the study
* Use of any medication or possession of any disease which, in the opinion of the investigator might interfere with the performance or interpretation of the study
* Laboratory tests changed (serum AST and ALT, alkaline phosphatase, urea and creatinine, total bilirubin and fractions)
* Patients with demonstrated hypercalcemia or evidence of toxicity of vitamin D
* Other conditions deemed reasonable by the medical investigator as to the disqualification of the individual from study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients will be selected from both sexes, healthy, between 18 and 65 years with a clinical diagnosis of chronic plaque psoriasis with PASI <20%, according to the criteria of inclusion and exclusion.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Schalka, Principal Investigator — Medcin Instituto da Pele Ltda